CLINICAL TRIAL: NCT05998655
Title: The Effect of Tele-Nursing Practices Based on Technological Competence Theory on Empowerment and Symptom Management in Breast Cancer Patients
Brief Title: Tele-nursing Practices Based on Technological Competence Theory in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Nisa YAVUZER BAYRAK, Research assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/787
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Female
Keywords: Tele-nursing; Technological Competence Theory; Breast Cancer; Cancer Empowerment; Symptom Management
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization will be made on a day-by-day basis due to the possibility of patients interacting in the outpatient clinic and waiting room during the research process. Before starting the research, a coin will be tossed to determine which group will be included on which day. If the money comes in summer, the patients who come on the first day will be taken to the experimental group, the patients who come on the second day will be taken to the control group. In the case of heads, the patients who come on the first day will be included in the control group, and the patients who come on the second day will be included in the experimental group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the data collection process, double-blindness will be ensured by not specifying which group the interviewer collects data from and which group the participants are from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In the research, tele-nursing practices and counseling based on the theory of technological competence will be provided to the experimental group.
  Interventions: Other: tele nursing
- control group (No Intervention): No attempt will be made on individuals in the control group during the research process

INTERVENTIONS:
Other: tele nursing — In the research, tele-nursing applications based on technological competence theory will be applied to the experimental group. In the content of the application, training, consultancy and follow-up will be made on breast cancer, the problems experienced in the treatment process of breast cancer, the most frequently experienced chemotherapy symptoms and management strategies. Technology knowledge will be based on the concepts of collaborative design and participant interaction. A five-week group training will be implemented once a week. The training will be applied to all the participants in the experimental group and will be held over "Google Meet". Educational program; pre-prepared powerpoint presentations, oral narration, discussion and group training will be made using e-booklets.
  Arms: experimental group

SUMMARY:
This research is a randomized controlled double-blind experimental study aiming to evaluate the effect of tele-nursing practices based on technological competence theory on empowerment status and symptom management self-efficacy in breast cancer patients. The research will be carried out between September 2023 and March 2024 with patients diagnosed with breast cancer, who are receiving chemotherapy on an active basis, registered in the Medical Oncology Polyclinic of Atatürk University Health Research and Application Center. The sample of the study will consist of 70 people, 35 of which are in the experimental group and 35 in the control group. Afterwards, approximately 11 weeks of tele-nursing practices, including training, counseling and tele-monitoring based on the theory of technological competence, will be given to the experimental group. While preparing the content of tele-nursing practices, national and international literature will be scanned. In line with the literature; Training, consultancy and follow-up will be provided on breast cancer, problems experienced in the treatment process of breast cancer, the most frequently experienced chemotherapy symptoms and management strategies. Before starting the training program, a training booklet will be distributed to the patients and shared as an e-booklet. Within the scope of the training program, a five-week training will be held once a week via "Google Meet". After the training program is completed, the counseling and telemonitoring process will begin. In this process, a previously prepared consultancy guide will be used. Counseling and telemonitoring will cover 2 chemotherapy cycles (approximately 6 weeks). Within the scope of the application, the entire experimental group will be individually phoned on the 7th day after receiving a chemotherapy course. Information about the individual conditions of the patients and the instant status changes regarding the symptoms will be obtained and their questions will be answered in line with the previously created counseling guide. Patients will be informed that at any time other than the specified days, the questions of the patients regarding the instantaneous situation changes will be answered. After the completion of the tele-nursing practices, post-test measurements will be made with the Cancer Empowerment Scale and the Chemotherapy Symptom Management in Breast Cancer-Self-efficacy Scale of the experimental and control groups, and the feedback of the patients in the experimental group regarding the implementation process will be received. No attempt will be made to the individuals in the control group during the research process.

Keywords: Tele-nursing, Technological Competence Theory, Breast Cancer, Cancer Empowerment, Symptom Management

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women globally. This situation is similar in our country and it is seen that one out of every four women diagnosed with cancer has breast cancer. Breast cancer is curable with 90% or higher survival rates, especially in the early stages of the disease. As treatment options, chemotherapy, radiotherapy, immunotherapy and surgical methods are used. These methods are applied in different combinations according to the stage and biological subtype of breast cancer. Chemotherapy, which is a frequently used treatment method in cancer treatment, is a systemic treatment method that aims to destroy cancer cells and stop their uncontrolled division. On the other hand, chemotherapy has many negative side effects and causes many physical and emotional symptoms. However, these symptoms can be prevented or reduced with effective treatment and nursing interventions. There are some skills expected from patients in order for the applied treatments and interventions to be effective. Among these skills are; Skills such as symptom management, lifestyle management or coping with the psychological effects of diseases can also be defined as self-management skills. At the stage of gaining these skills, the concept of empowerment of cancer patients emerges. Cancer enhancement; It is a process in which patients specialize in treatment, care and diseases. Empowerment also provides access to high-quality and appropriate care, improved quality of life, better interaction with healthcare professionals, better response to treatment, prevention of complications, and positive attitude towards illness. An empowered patient is an informed patient who takes responsibility for his or her health as much as possible. The vast majority of patients receiving neoadjuvant chemotherapy receive chemotherapy on an outpatient basis. This causes symptoms to be self-managed at home for a long period of time. On the other hand, breast cancer is subjective and every person experiences it differently, and responses to the disease and treatment differ individually. For this reason, it is important to provide individual counseling and professional support in the process of coping with the side effects of chemotherapy. With the development of technology, it is necessary to ensure a harmonious coexistence between nursing care and technology. The theory of 'Technological Competence in Nursing Care', which was developed based on these requirements, is one of the relatively new nursing theories and models. According to the theory, the aim of technological competence in nursing; accepting the patient as a focal point of nursing and benefiting from various technological tools in nursing interventions and defining the individual. According to the International Nurses Association (ICN), tele-nursing; According to the American Nurses Association (ANA), it is defined as the use of communication technologies in nursing to improve patient care, and nursing practices such as obtaining information about the health status of patients, providing care, and patient education by using communication technologies. In this context, tele-nursing is compatible with the concepts and assumptions of the technological competence theory. Women with breast cancer experience numerous physical, psycho-social and sexual complications arising from the disease and treatment methods, and many roles of women are damaged due to the disease. Symptoms experienced during and after chemotherapy treatment negatively affect the patient's empowerment and symptom management. In this process, patients often refer to internet resources to get information about the disease and the symptoms experienced. However, there are doubts about the accuracy of the information obtained and the level of evidence. In a study conducted with people with breast cancer, it was determined that sometimes the information obtained from different internet sources is incomplete or even inconsistent, causing confusion. In another study, it was determined that people with breast cancer think that empowerment is important during the illness and that empowerment issues should include knowledge, beliefs and skills. In this context, it is thought that tele-nursing practices based on technological competence theory will increase empowerment in breast cancer patients and benefit the symptom management self-efficacy. Breast cancer patients are involved in a long and difficult life process from diagnosis. After the shock process of being diagnosed with cancer, it is necessary to be involved in a treatment process quickly. Due to some side effects experienced during the treatment process, they experience some physical, psychological, sexual, occupational and many more problems. While these problems may improve from time to time, there may also be exacerbations. In fact, some adaptation problems may be experienced in the process and patients may even consider stopping the treatment due to the symptoms they experience. In this context, individual counseling and professional support to be provided to patients is very important for the effectiveness of the treatment, which must be continued in a long and difficult process. In a systematic review study evaluating the effectiveness of nursing interventions for breast cancer patients according to the literature, it was determined that nurse-led teaching, guidance, counseling and case management interventions were effective for symptom management. On the other hand, it has been found that the symptom management of patients is poorly controlled despite various guidance in different studies. For this reason, new studies with different models are required in order to provide management skills more powerfully. The concept of patient empowerment is growing in importance in health-related research, and studies show that empowerment improves care outcomes and increases patient satisfaction in those with chronic illness. Thanks to the advances in early diagnosis and treatment technology of breast cancer, survival rates have increased and it has started to be seen as a chronic disease. In most of the studies on the subject, it is seen that augmentation-related interventions are effective, but generally work with breast cancer survivors. However, the fact that the population defined as breast cancer survivors, that is, who completed the breast cancer treatment process, has more experience compared to their newly diagnosed peers and partially knew what to do and how to do it, suggests that they may need an information tool less. In this context, breast cancer patients should be informed about their disease throughout their lives and during the chemotherapy process in order to strengthen their symptom management skills while their treatment continues. When the literature is evaluated, it is seen that information studies conducted with breast cancer patients receiving chemotherapy are generally conducted in the outpatient chemotherapy unit, even while the patient is receiving chemotherapy drugs. In this process, it is thought that breast cancer patients are in the hospital environment and in a crowded environment, they experience the early side effects of the treatment intensely, they have difficulty in managing the symptoms they experience at home and in reaching adequate counseling and support when they need it, and for this reason, they cannot fully benefit from the information/education studies. For this reason, it is expected that informing the patient with tele-nursing practices while the patient is at home during the periods when the patients feel better and the early side effects of chemotherapy decrease, and until the next cure treatment will contribute both in terms of the patient and the skill development expected from the patient. There are some studies evaluating the effects of web-based and mobile application interventions in breast cancer patients. It has been found that the applications made in these studies provide clinical improvement in conditions such as symptom control and management, self-management behaviors, functional exercise compliance, quality of life and drug compliance. No study has been found that evaluates the effects of tele-nursing practice, which is based on technological competence theory and focuses on self-efficacy, especially on empowerment and symptom management, in breast cancer patients receiving neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer I., II. or III. in phase
* Without organ metastases
* Those who have not been diagnosed with any other cancer other than breast cancer
* Literate
* Receiving neoadjuvant chemotherapy
* Received at least 1 course of chemotherapy
* Those who does not have hearing and speech problems that will prevent talking on the phone
* Capable of using a smartphone
* Does not have any psychiatric problems that reduce the ability to understand
* Who volunteered to participate in the research

Exclusion Criteria:

* With stage 4 breast cancer
* Organ metastases
* Those who have been diagnosed with a cancer other than breast cancer
* iliterate
* Cannot communicate verbally
* Unable to use a smartphone
* No internet connection or online access
* Who refused to participate in the research

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer in women
Enrollment: 70 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Cancer Empowerment Scale | 11 week
  n 2013, Van den Berg et al. The 'Cancer Empowerment Scale', developed ., is a 40-item scale created to understand the empowerment of patients in coping with their diseases during their illness. It was adapted into Turkish by Karabulutlu, et al., (2021) and consists of 4 sub-dimensions: personal power, social support, health care and community. The total Cronbach's alpha coefficient of the scale is 0.93, and the increase in the total score and the mean score of the sub-dimensions indicates that the patients become stronger in this disease process.
Chemotherapy Symptom Management in Breast Cancer-Self-Efficacy Scale | 11 week
  iang et al. (2015) Chemotherapy Symptom Management-Self-Efficacy Scale was developed to evaluate symptom management and self-efficacy in breast cancer patients undergoing chemotherapy. The scale, which was adapted into Turkish by Semiz D., and Sağlam R. (2018), consists of 3 sub-dimensions and 27 items: problem-solving skills, management of chemotherapy-related symptoms, and management of emotional-interpersonal problems. Items are scored on a 0-10 point likert scale (0 = not at all sure, 10 = very sure). The total score is obtained by adding the digits of each answer from the scale. The score for the entire scale ranges from 0 to 270. When calculating the scores on the scale items, a high score indicates that the person's perceived self-efficacy in managing symptoms is high

CONTACTS AND LOCATIONS:
Overall Officials: Nisa YAVUZER BAYRAK, Principal Investigator — Ataturk University; Elanur YILMAZ KARABULUTLU, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)